CLINICAL TRIAL: NCT00769704
Title: A Randomized Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of Treatment With OncoVEX^GM-CSF Compared to Subcutaneously Administered GM-CSF in Melanoma Patients With Unresectable Stage IIIb, IIIc and IV Disease
Brief Title: Efficacy and Safety Study of Talimogene Laherparepvec Compared to Granulocyte Macrophage Colony Stimulating Factor (GM-CSF) in Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioVex Limited (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 005/05; 20110263 (Other: Sponsor); 2008-006140-20 (EudraCT Number)
Record Dates: First submitted 2008-10-07; First posted 2008-10-09 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-06

CONDITIONS: Melanoma
Keywords: Melanoma; OncoVEX^GM-CSF; GM-CSF; Stage IIIb, IIIc and IV Disease; oncolytic; OncoVex; T-Vec; talimogene laherparepvec
MeSH Terms: conditions — Melanoma | interventions — talimogene laherparepvec; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GM-CSF (Active Comparator): Granulocyte macrophage colony-stimulating factor (GM-CSF) was administered at a dose of 125 μg/m²/day subcutaneously for 14 days, followed by a 14-day rest period for 24 weeks. Participants could continue treatment until clinically relevant disease progression, intolerability, withdrawal of consent, complete remission, or lack of response by 12 months, for a maximum of 18 months.
  Interventions: Biological: GM-CSF
- Talimogene Laherparepvec (Experimental): Participants received talimogene laherparepvec on Days 1 and 15 of each 28-day cycle for 24 weeks. The initial dose of talimogene laherparepvec was at a concentration of 10⁶ plaque forming units (PFU)/mL, injected into 1 or more skin, subcutaneous or nodal tumors. Subsequent doses began at least 3 weeks after the first dose and consisted of talimogene laherparepvec at a concentration of 10⁸ PFU/mL. Participants could continue treatment until clinically relevant disease progression, intolerability, withdrawal of consent, complete remission, lack of response by 12 months, or disappearance of all injectable lesions, for a maximum of 18 months.
  Interventions: Biological: Talimogene laherparepvec

INTERVENTIONS:
Biological: Talimogene laherparepvec — Up to 4 mL of 10⁸ pfu/mL/per intratumoral injection
  Other Names: OncoVEX^GM-CSF; IMLYGIC™
  Arms: Talimogene Laherparepvec
Biological: GM-CSF — 125 µg/m² subcutaneous injection
  Other Names: Leukine; Sargramostim
  Arms: GM-CSF

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of treatment with talimogene laherparepvec compared to subcutaneously administered GM-CSF in patients with unresectable Stage IIIb, IIIc and Stage IV melanoma. The efficacy endpoints of the study aim to demonstrate overall clinical benefit for patients treated with talimogene laherparepvec as compared to GM-CSF.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age ≥ 18 years
* Stage IIIb, IIIc or stage IV disease that is not surgically resectable
* Injectable disease (i.e. suitable for direct injection or through the use of ultrasound guidance)
* At least 1 injectable cutaneous, subcutaneous or nodal melanoma lesion >= 10 mm in longest diameter or, multiple injectable melanoma lesions which in aggregate have a longest diameter of >= 10 mm
* Serum lactate dehydrogenase (LDH) levels less than 1.5 x upper limit of normal (ULN)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Prolongation in International Normalized Ratio (INR), Prothrombin Time (PT), and Partial Thromboplastin Time (PTT) when the result is from therapeutic anticoagulation treatment are permitted for patients whose injectable lesions are cutaneous and/or subcutaneous such that direct pressure could be applied in the event of excessive bleeding

Exclusion Criteria:

* Clinically active cerebral or any bone metastases. Patients with up to 3 (neurological performance status of 0) cerebral metastases may be enrolled, provided that all lesions have been adequately treated with stereotactic radiation therapy, craniotomy, gammaknife therapy, with no evidence of progression, and have not required steroids, for at least two (2) months prior to randomization
* Greater than 3 visceral metastases (this does not include lung metastases or nodal metastases associated with visceral organs). For patients with < 3 visceral metastases, no lesion > 3 cm, and liver lesions must meet Response Evaluation Criteria In Solid Tumors (RECIST) criteria for stable disease for at least 1 month prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 437 (Actual)
Dates: Start 2009-04; Primary Completion 2013-02 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (83):
- United States (57):
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego, Moores Cancer Center, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - San Francisco Oncology Associates, San Francisco, California
  - Northern California Melanoma Center, St. Mary's Medical Center, San Francisco, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Redwood Regional Medical Group Inc, North Bay Melanoma Program, Sebastopol, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Baptist Cancer Institute, Jacksonville, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - University of Miami, Miami, Florida
  - Mount Sinai Medical Center CCOP, Miami Beach, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Cancer Care Center at Lutheran General Hospital, Park Ridge, Illinois
  - Indiana University, Indianapolis, Indiana
  - Investigative Clinical Research of Indiana, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Hubert H Humphrey Cancer Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Kansas City Cancer Center, Kansas City, Missouri
  - St. Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Mountainside Hospital, Morristown, New Jersey
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia Medical University, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of North Carolina At Chapel Hill School of Medicine, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Barrett Cancer Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Taussig Cancer Center, Cleveland, Ohio
  - Earle A Chiles Research Institute, Providence Cancer Center, Portland, Oregon
  - St Luke's Hospital & Health Network, Bethlehem, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Institute for Translational Oncology Research, Greenville, South Carolina
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Texas Cancer Center, Abilene, Abilene, Texas
  - Mary Crowley Medical Research Center, Dallas, Texas
  - University of Texas - MD Anderson, Houston, Texas
  - Texas Oncology, Allison Cancer Center, Midland, Texas
  - Intermountain Medical Center, Murray, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Salem, Virginia
  - Aurora/St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- South Africa (10):
  - GVI Oncology, Port Elizabeth, Eastern Cape
  - Dr. Fourie & Bonnet, Bloemfontein, Free State
  - Medical Oncology Centre of Rosebank, Johannesburg, Gauteng
  - Wits Donald Gordon Clinical Trial Site, Parktown, Guateng
  - University of Pretoria, Pretoria, Guateng
  - Mary Potter Oncology Centre, Pretoria, Guateng
  - Hopelands Cancer Centre, Pietermaritzburg, KwaZulu-Natal
  - Wilgers Oncology Center, Hatfield, Pretoria
  - GVI Onocology Clinical Trials Unit, Cape Town, Western Cape
  - GVI Oncology Centre, Cape Town, Western Cape
- United Kingdom (13):
  - University of Birmingham, Birmingham
  - Addenbrookes Hospital, Cambridge
  - Broomfield Hospital, Chelmsford
  - St. James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Royal Free Hospital, London
  - St. George's University of London, London
  - Royal Marsden Hospital, London
  - Clatterbridge Centre for Oncology, Metropolitan Borough of Wirral
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Southampton General Hospital, Southampton

REFERENCES:
- [Result] Andtbacka RH, Kaufman HL, Collichio F, Amatruda T, Senzer N, Chesney J, Delman KA, Spitler LE, Puzanov I, Agarwala SS, Milhem M, Cranmer L, Curti B, Lewis K, Ross M, Guthrie T, Linette GP, Daniels GA, Harrington K, Middleton MR, Miller WH Jr, Zager JS, Ye Y, Yao B, Li A, Doleman S, VanderWalde A, Gansert J, Coffin RS. Talimogene Laherparepvec Improves Durable Response Rate in Patients With Advanced Melanoma. J Clin Oncol. 2015 Sep 1;33(25):2780-8. doi: 10.1200/JCO.2014.58.3377. Epub 2015 May 26. PMID 26014293
- [Derived] Andtbacka RHI, Collichio F, Harrington KJ, Middleton MR, Downey G, Ӧhrling K, Kaufman HL. Final analyses of OPTiM: a randomized phase III trial of talimogene laherparepvec versus granulocyte-macrophage colony-stimulating factor in unresectable stage III-IV melanoma. J Immunother Cancer. 2019 Jun 6;7(1):145. doi: 10.1186/s40425-019-0623-z. PMID 31171039
- [Derived] Kaufman HL, Andtbacka RHI, Collichio FA, Wolf M, Zhao Z, Shilkrut M, Puzanov I, Ross M. Durable response rate as an endpoint in cancer immunotherapy: insights from oncolytic virus clinical trials. J Immunother Cancer. 2017 Sep 19;5(1):72. doi: 10.1186/s40425-017-0276-8. PMID 28923101

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were adults with histologically confirmed, not surgically resectable, stage IIIB - IV melanoma suitable for direct or ultrasound-guided injection.
  Among those randomized, the first patient enrolled 29 April 2009 and last patient enrolled 8 June 2011.
  1 patient randomized 3 times is counted once under talimogene laherparepvec.
Pre-assignment Details: Patients were assigned at a 2:1 ratio using central random assignment to receive intralesional talimogene laherparepvec or subcutaneous granulocyte macrophage colony-stimulating factor (GM-CSF). Randomization was stratified by site of first recurrence, presence of liver metastases, disease stage, and prior nonadjuvant systemic treatment.
Groups:
- GM-CSF: Granulocyte macrophage colony-stimulating factor (GM-CSF) was administered at a dose of 125 μg/m²/day subcutaneously for 14 days in 28-day cycles for 24 weeks. Participants could continue treatment until clinically relevant disease progression, intolerability, withdrawal of consent, complete remission, or lack of response by 12 months, for a maximum of 18 months.
Period: Overall Study
Arm/Group | GM-CSF | Talimogene Laherparepvec
Started | 141 | 296
Intent-to-treat Population | 141 (All participants who were randomized once to study treatment) | 295 (Participants who were randomized once to study treatment; excludes 1 participant randomized 3 times)
Received Treatment | 127 | 292
Completed | 30 | 97
Not Completed | 111 | 199
Not completed — Lost to Follow-up | 3 | 2
Not completed — Death | 95 | 190
Not completed — Withdrawal by Subject | 12 | 5
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- GM-CSF: GM-CSF was administered at a dose of 125 μg/m²/day subcutaneously for 14 days in 28-day cycles for 24 weeks. Participants could continue treatment until clinically relevant disease progression, intolerability, withdrawal of consent, complete remission, or lack of response by 12 months, for a maximum of 18 months.
- Talimogene Laherparepvec: Participants received talimogene laherparepvec on Days 1 and 15 of each 28-day cycle for 24 weeks. The initial dose was at a concentration of 10⁶ PFU/mL, injected into 1 or more skin, subcutaneous or nodal tumors. Subsequent doses began at least 3 weeks after the first dose and consisted of talimogene laherparepvec at a concentration of 10⁸ PFU/mL. Participants could continue treatment until clinically relevant disease progression, intolerability, withdrawal of consent, complete remission, lack of response by 12 months, or disappearance of all injectable lesions, for a maximum of 18 months.
- Total: Total of all reporting groups
Arm/Group | GM-CSF | Talimogene Laherparepvec | Total
Number analyzed (Participants) | 141 | 296 | 437
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.92 (14.13) | 63.07 (13.68) | 63.03 (13.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 123 | 187
  Male | 77 | 173 | 250
Race/Ethnicity, Customized [Number; unit: participants]
  White | 138 | 290 | 428
  Black | 2 | 1 | 3
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Other | 1 | 3 | 4
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Scale used to assess how a patient's disease is progressing, how the disease affects the daily living abilities of the patient: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory, able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self care, confined to a bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  participants
    0 | 97 | 210 | 307
    1 | 32 | 82 | 114
    Missing | 12 | 4 | 16
Tumor, Node, Metastasis (TNM) Disease Stage [Number; unit: participants] — Stage IIIB: Ulcerated lesion and 1 lymph node or 2-3 nodes with micrometastasis, or any-depth lesion with no ulceration, and 1 lymph node or 2-3 nodes with macrometastasis; Stage IIIC: Ulcerated lesion and 1 lymph node with macrometastasis; 2-3 nodes with macrometastasis or ≥4 metastatic lymph nodes, matted lymph nodes, or in-transit met(s)/satellite(s); Stage IV: M1a: Spread to skin, subcutaneous tissue, or lymph nodes; normal lactate dehydrogenase (LDH) level; M1b: Spread to lungs, normal LDH; M1c: Spread to all other visceral organs, normal LDH or any distant disease with elevated LDH.
  participants
    Stage IIIB | 12 | 22 | 34
    Stage IIIC | 31 | 66 | 97
    Stage IV M1a | 43 | 76 | 119
    Stage IV M1b | 26 | 64 | 90
    Stage IV M1c | 29 | 67 | 96
    Missing | 0 | 1 | 1
Line of Therapy [Number; unit: participants]
  First Line | 65 | 138 | 203
  Second Line or Greater | 76 | 158 | 234

OUTCOME MEASURES:

1. Primary Outcome: Durable Response Rate
Description: Durable response rate was defined as the percentage of participants with a complete response (CR) or partial response (PR) maintained continuously for at least 6 months from the time the objective response was first observed and initiating within 12 months of starting therapy as assessed by the Endpoint Assessment Committee (EAC). This reflects all new sites of disease as well as disease sites identified at baseline.
  Disease assessments were performed at the beginning of each treatment cycle in accordance with modified World Health Organization criteria.
  CR: Disappearance of all clinical evidence of tumor (both measurable and non-measurable but evaluable disease); PR: ≥ 50% reduction in the sum of the products of the perpendicular diameters of all measurable tumors at the time of assessment as compared to baseline.
Time Frame: From randomization until the data cut-off date of 21 December 2012; median follow-up time was 20 months.
Population: Intent-to-treat population (all participants randomized to receive study treatment), excluding one participant who was randomized three times.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GM-CSF | Talimogene Laherparepvec
Number analyzed (Participants) | 141 | 295
percentage of participants | 2.1 [0.0 to 4.5] | 16.3 [12.1 to 20.5]
Statistical Analysis 1: Comparison: GM-CSF vs Talimogene Laherparepvec; The null hypothesis was that there was no difference in the durable response rate between the talimogene laherparepvec and control arms. Study success was defined as the rejection of this hypothesis such that talimogene laherparepvec was found to be superior to GM-CSF using the 2-sided Fisher's exact test, with a p-value of ≤ 0.0488; Test type: Superiority or Other; p < 0.0001, Fisher Exact; Treatment Difference = 14.1, 95% CI 2-sided [9.3 to 19.0]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of randomization to the date of death from any cause. Overall survival time was censored at the last date the patient was known to be alive when the confirmation of death was absent or unknown. Participants were censored at the date of randomization if no additional follow-up data were obtained.
Time Frame: From randomization until the first 290 survival events had occurred (data cut-off date of 31 March 2014); median time on follow-up was 44 months.
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GM-CSF | Talimogene Laherparepvec
Number analyzed (Participants) | 141 | 295
months | 18.9 [16.0 to 23.7] | 23.3 [19.5 to 29.6]
Statistical Analysis 1: Comparison: GM-CSF vs Talimogene Laherparepvec; The primary method for analysis of overall survival was an unadjusted log-rank test. Testing of overall survival was conditional on a statistically significance difference in the primary endpoint of durable response. Success was defined as a p-value ≤ 0.05; Test type: Superiority or Other; p = 0.0511, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.62 to 1.00] — The hazard ratio was obtained from the unadjusted Cox Proportional Hazard Model. A hazard ratio < 1.0 indicates a lower average death rate and a longer overall survival for talimogene laherparepvec relative to GM-CSF

3. Secondary Outcome: Objective Response Rate
Description: Objective response rate was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) assessed by the Endpoint Assessment Committee (EAC). Best overall response for a patient is the best overall response observed across all time points.
  Disease assessments were performed at the beginning of each treatment cycle and assessed in accordance with modified World Health Organization criteria.
  CR: Disappearance of all clinical evidence of tumor (both measurable and non-measurable but evaluable disease); PR: ≥ 50% reduction in the sum of the products of the perpendicular diameters of all measurable tumors at the time of assessment as compared to baseline.
Time Frame: From randomization until the data cut-off date of 21 December 2012; median follow-up time was 20 months.
Population: Intent-to-treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GM-CSF | Talimogene Laherparepvec
Number analyzed (Participants) | 141 | 295
percentage of participants | 5.7 [1.9 to 9.5] | 26.4 [21.4 to 31.5]
Statistical Analysis 1: Comparison: GM-CSF vs Talimogene Laherparepvec; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Descriptive; Treatment Difference = 20.8, 95% CI 2-sided [14.4 to 27.1]

4. Secondary Outcome: Duration of Response
Description: The duration of response is defined as the longest individual period from entering response (CR or PR as assessed by the EAC) to the first documented evidence of the patient no longer meeting the criteria for being in response or death, whichever is earlier. Responses were censored at the last assessment showing response.
Time Frame: From randomization until the data cut-off date of 21 December 2012; median follow-up time was 20 months.
Population: Participants with an objective response (CR or PR) per EAC assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GM-CSF | Talimogene Laherparepvec
Number analyzed (Participants) | 8 | 78
months | 2.8 [1.2 to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: GM-CSF vs Talimogene Laherparepvec; Test type: Superiority or Other; p = 0.0868, Log Rank — Descriptive; Hazard Ratio (HR) = 0.40, 95% CI 2-sided [0.14 to 1.18] — The hazard ratio was obtained from the unadjusted Cox Proportional Hazard Model. A hazard ratio < 1.0 indicates a longer average duration of response for talimogene laherparepvec relative to GM-CSF

5. Secondary Outcome: Response Onset
Description: Response onset is defined as the time from the date of randomization to the date of the first documented evidence of response (CR or PR) per EAC assessment.
Time Frame: From randomization until the data cut-off date of 21 December 2012; median follow-up time was 20 months.
Population: Participants with an objective response (CR or PR) per EAC assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GM-CSF | Talimogene Laherparepvec
Number analyzed (Participants) | 8 | 78
months | 3.7 [1.9 to 5.6] | 4.1 [3.8 to 5.4]
Statistical Analysis 1: Comparison: GM-CSF vs Talimogene Laherparepvec; Test type: Superiority or Other; p = 0.2020, Log Rank — Descriptive; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.30 to 1.30] — The hazard ratio was obtained from the unadjusted Cox Proportional Hazard Model. A hazard ratio > 1.0 indicates a a higher average response onset rate for talimogene laherparepvec relative to GM-CSF

6. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was assessed by the investigator, and calculated from randomization until the first clinically relevant disease progression where there is no response achieved after the progression, or until death if no such progression occurs. Participants who did not have clinically relevant progression or did not die were censored at the time of the their last tumor assessment. Participants who withdrew from treatment due to a clinically unacceptable toxicity were not considered as an event in the analysis.
  Progressive disease (PD) is defined as a ≥ 25% increase in the sum of the products of the perpendicular diameters of all measurable tumors since baseline, or the unequivocal appearance of a new tumor since the last response assessment time point.
  Clinically relevant progressive disease is PD that is associated with a decline in performance status and/or in the opinion of the investigator the patient requires alternative therapy.
Time Frame: From randomization until the data cut-off date of 21 December 2012; median follow-up time was 20 months.
Population: Intent to treat population
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Talimogene Laherparepvec: Participants received talimogene laherparepvec on Days 1 and 15 of each 28-day cycle for 24 weeks. The initial dose was at a concentration of 10⁶ plaque forming units (PFU)/mL, injected into 1 or more skin, subcutaneous or nodal tumors. Subsequent doses began at least 3 weeks after the first dose and consisted of talimogene laherparepvec at a concentration of 10⁸ PFU/mL. Participants could continue treatment until clinically relevant disease progression, intolerability, withdrawal of consent, complete remission, lack of response by 12 months, or disappearance of all injectable lesions, for a maximum of 18 months.
Arm/Group | GM-CSF | Talimogene Laherparepvec
Number analyzed (Participants) | 141 | 295
months | 2.9 [2.8 to 4.0] | 8.2 [6.5 to 9.9]
Statistical Analysis 1: Comparison: GM-CSF vs Talimogene Laherparepvec; Test type: Superiority or Other; p < 0.0001, Log Rank — Descriptive; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.32 to 0.54] — The hazard ratio was obtained from the unadjusted Cox Proportional Hazard Model. A hazard ratio < 1.0 indicates a longer average time to treatment failure for talimogene laherparepvec relative to GM-CSF

7. Secondary Outcome: Response Interval
Description: Response interval is defined as the interval between the date of randomization and the date of the last documented evidence of response (CR or PR as assessed by the Investigator) prior to any new anti-cancer therapy. Response Interval post response onset was censored if a patient was still in response at the last observation.
Time Frame: From randomization until the data cut-off date of 21 December 2012; median follow-up time was 20 months.
Population: Participants with an objective response (CR or PR) per Investigator assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | GM-CSF | Talimogene Laherparepvec
Number analyzed (Participants) | 9 | 91
months | 7.5 [1.9 to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: GM-CSF vs Talimogene Laherparepvec; Test type: Superiority or Other; p = 0.0050, Log Rank — Descriptive; Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.13 to 0.73] — The hazard ratio was obtained from the unadjusted Cox Proportional Hazard Model. A hazard ratio < 1.0 indicates a longer response interval for talimogene laherparepvec relative to GM-CSF

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 30 days after the last dose; Median duration of treatment was 10 weeks (range 0.6 to 72 weeks) in GM-CSF group and 23 weeks (range 0.1 to 78.9 weeks) in the talimogene laherparepvec group.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | GM-CSF | Talimogene Laherparepvec
Serious Adverse Events (participants affected / at risk) | 17/127 | 75/292
Other Adverse Events (participants affected / at risk) | 112/127 | 282/292
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GM-CSF (N=127) | Talimogene Laherparepvec (N=292)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Intussusception (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Disease progression (General disorders) | 2 | 9
Influenza like illness (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 5
Cellulitis (Infections and infestations) | 1 | 7
Gastroenteritis (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Radiation associated pain (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Wound decomposition (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Brain oedema (Nervous system disorders) | 0 | 1
Central nervous system lesion (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 3
Convulsion (Nervous system disorders) | 0 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Pneumocephalus (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 2
Glomerulonephritis (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal papillary necrosis (Renal and urinary disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GM-CSF (N=127) | Talimogene Laherparepvec (N=292)
Anaemia (Blood and lymphatic system disorders) | 2 | 15
Abdominal pain (Gastrointestinal disorders) | 3 | 26
Constipation (Gastrointestinal disorders) | 8 | 34
Diarrhoea (Gastrointestinal disorders) | 14 | 55
Dyspepsia (Gastrointestinal disorders) | 8 | 15
Nausea (Gastrointestinal disorders) | 25 | 104
Vomiting (Gastrointestinal disorders) | 12 | 61
Chills (General disorders) | 11 | 141
Fatigue (General disorders) | 46 | 147
Influenza like illness (General disorders) | 19 | 88
Injection site erythema (General disorders) | 33 | 15
Injection site pain (General disorders) | 8 | 81
Injection site pruritus (General disorders) | 21 | 5
Injection site reaction (General disorders) | 12 | 9
Injection site swelling (General disorders) | 8 | 10
Oedema peripheral (General disorders) | 12 | 34
Pain (General disorders) | 13 | 47
Pyrexia (General disorders) | 11 | 121
Upper respiratory tract infection (Infections and infestations) | 8 | 29
Weight decreased (Investigations) | 1 | 17
Decreased appetite (Metabolism and nutrition disorders) | 14 | 30
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 50
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 27
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 51
Neck pain (Musculoskeletal and connective tissue disorders) | 7 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 48
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 19
Dizziness (Nervous system disorders) | 4 | 28
Headache (Nervous system disorders) | 12 | 55
Anxiety (Psychiatric disorders) | 2 | 19
Depression (Psychiatric disorders) | 3 | 15
Insomnia (Psychiatric disorders) | 6 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 31
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 17
Erythema (Skin and subcutaneous tissue disorders) | 9 | 21
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9 | 23
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 28
Rash (Skin and subcutaneous tissue disorders) | 10 | 26
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.